CLINICAL TRIAL: NCT04100629
Title: The Impact of a Digital Support Intervention on Stress, Resiliency, Perceived Social Support, and Intention to Leave Among Newly Licensed Nurses: A Randomized Controlled Trial
Brief Title: Digital Support Intervention on Newly Licensed Nurses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment (and due to pandemic)
Sponsor: Duquesne University (Other)
Collaborators: West Penn Allegheny Health System (Other); University of California, San Diego (Other); El Centro Medical Center (Unknown); Pioneers Hospital (Unknown)
Responsible Party: Principal Investigator, Lisa A Concilio, Principle Investigator, Duquesne University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/06/10
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Stress; Job Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: A prospective, RCT design with an experimental and control group is proposed for this study to determine if a digital support intervention impacts Newly Licensed Nurses' stress, resiliency, perceived sense of support, and Intention To Leave their current jobs.
Who Masked: Participant
Masking Description: participants' unique numeric identifiers will be separated into two groups by the random generator with the exception of male participants. To enhance similarity among the control and experimental groups, male participants will be evenly distributed between groups (every other male, in sequential order of data collection, will be placed into each group) and not randomized (Polit & Beck, 2017).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will receive medical facts and are not meant to support newly licensed nurses and are not known to affect stress, resilience, perceived social support, or Intention To Leave one's job.
  Interventions: Behavioral: digital support: text messages
- Experimental Group (Experimental): Texts sent to the experimental group will be based on nurturant support messages and are intended to decrease stress, Intention To Leave, increase resilience, and perceived sense of support.
  Interventions: Behavioral: digital support: text messages

INTERVENTIONS:
Behavioral: digital support: text messages — In this study, the text messages are intended to be one-directional, from the PI to the participant. Participants are not expected to reply. If participants reply to any of the text messages, the PI will screen the content and only reply if it is a question regarding the study or a request to seek counseling. Additionally, participants will be instructed by the PI to access their Smartphones to read texts while on a break, after their shift, or when not at work; participants will be instructed to not use Smartphones to read texts while working. A series of four text messages will be sent to all study participants (experimental and control groups) by the PI every Monday, Wednesday, Friday, and Saturday (M, W, F, S) at 1pm for six weeks, for a total of 24 different texts for each group.
  Other Names: text messages

SUMMARY:
Brief Description of the Study: Text messages will be sent to participants and responses will be surveyed to ascertain if using a social, digital intervention can influence NLNs' (newly licensed nurses') stress, resiliency, perceived sense of social support, and/or the intention to stay at current jobs. Newly licensed nurses (within their first year of hire) will be asked to participate. A series of four text messages will be sent to all study participants (experimental and control groups) by the PI every Monday, Wednesday, Friday, and Saturday (M, W, F, S) at 1pm for six weeks, for a total of 24 different texts for each group. Participants will fill out surveys before the study begins, at week 3 and at the end of the study (week 6).The control group will receive medical facts. Texts sent to the experimental group will be based on SSBC nurturant support messages and are intended to decrease stress intention to leave (ITL), increase resilience, and perceived sense of support. The SSBC nurturant support texts are comprised of three themes of support: emotional, network, and esteem. The experimental group's supportive text messages were created by the PI and require content validation. A gatekeeper at your facility will be asked to send an email to "Experts" (MSN educators) and ask them to complete the validation survey using a Qualtrics Survey Platform then the PI will place ratings into a table and calculate the results. There are 3 other facilities enrolled in this study: University California, San Diego, El Centro Medical Center, and Pioneer Hospital (all located in southern California).

DETAILED DESCRIPTION:
The purpose of this randomized control study (RCT) is to determine the impact of a 6-week digital support intervention (text messaging) on NLNs' levels of stress, resiliency, perceived social support, and ITL (intention to leave) their current jobs. The long-term objective is to examine if a 6-week digital support intervention impacts NLNs' (newly licensed nurses') ITL during the first year of hire. The central hypothesis is that a digital support intervention plays a critical role in NLNs' levels of stress, resilience, perceived sense of social support, and ITL their current jobs. In order to be included in this proposed study, participants must agree to not use their Smartphones while providing direct patient care but may access text messages while in designated break areas or when off duty.

Research Questions: RQ1: What is the effect of a digital support intervention upon NLNs' stress? RQ2: What is the effect of a digital support intervention upon NLNs' resiliency? RQ3: What is the effect of a digital support intervention upon NLNs' perceived social support? RQ4: What is the effect of a digital support intervention upon NLNs' ITL their first jobs during their first year of hire?

Design (Description of research plan, intervention(s) and time frame): A prospective, RCT design with an experimental and control group is proposed for this study to determine if a digital support intervention impacts NLNs' stress, resiliency, perceived sense of support, and Intention to Leave.

ELIGIBILITY:
Inclusion Criteria:

* Newly Licensed Nurses,
* ages 19-37 years,
* proficient in English,
* working in an acute care facility as a RN during the first year of hire,
* have a working personal Smartphone,
* have the ability to send and receive text messages,
* have an active and working personal email account, and
* be willing to participate for six weeks,
* complete a demographic survey before the study, survey instruments at 3 weeks, 6 weeks, and at the conclusion of the study
* agree to not use or carry their Smartphone while performing direct patient care and
* assume any data charges for text messages, if incurred.

Exclusion Criteria:

* Newly Licensed Nurses who have worked in the role of a RN on another floor or
* NLNs who have worked as an RN at another organization, or
* NLNs not 19-37 years of age.

Ages: 19 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Reported levels of perceived stress will change; predicted to decrease. | prior to intervention, 3 weeks, and 6 weeks
  The Perceived Stress Scale (PSS) will be used to measure stress (Cohen, Kamarck, & Mermelstein, 1983). Participant stress will measured prior to intervention, at 3 weeks, and 6 weeks. It is a 10-item, Likert-type scale with five points. Scores are obtained by using the item responses that range from 0 to 4 (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often) with items 4, 5, 7, and 8 reversely scored. The summed scores of the PSS will be used for one of the dependent variables and will be discussed further as a key variable. Participants will be asked to think about their current work situation when answering survey questions. The possible range of scores, after adding all points, will range from 0 to 40, with higher scores signifying greater perceived stress.
Report levels of resiliency will change; predicted to increase. | prior to intervention, 3 weeks, and 6 weeks
  The Connor-Davidson Resiliency Scale (CD-RISC-25) will be used to measure resiliency (Connor & Davidson, 2003). Participant resilience will measured prior to intervention, at 3 weeks, and 6 weeks. The CD-RISC-25 is a 25-item self-report scale that uses a five-point Likert-type scale ranging from 0 (not true at all) to 4 (true nearly all the time). Total scores, ranging from 0-100, assess resilience and a score of 100 denotes the highest level of resiliency; the tool takes 5-10 minutes to complete (CD RISC, 2011). The summed scores of the CD-RISC 25 will be used for one of the dependent variables and will be discussed further as a key variable.
Reported levels of participants Sense of Support will change; predicted to increase. | prior to intervention, 3 weeks, and 6 weeks
  The Social Support Scale (SSS) will be used to measure perceived social support scores (Dolbier & Steinhardt, 2000). Participant perceived social support will measured prior to intervention, at 3 weeks, and 6 weeks. Respondents answer 21 items on a 4-option Likert-type scale labeled between 0 (not true at all) to 3 (completely true) (Dolbier & Steinhardt, 2000) and will take 20-25 minutes to complete (Versta, 2011). The summed scores of the SSS will be used for one of the dependent variables and will be discussed further as a key variable.
Intentions to Leave current job will change; predicted to decrease. | 6 weeks
  An "Intention to Leave," investigator designed survey will be used to measure the participants' Intention to Leave their current jobs. Participant intention to leave their current job will measured at 6 weeks. Participants will be asked what percentage, if any, represents their ITL their current position and also what percentage represents their ITL to leave their current organization.

CONTACTS AND LOCATIONS:
Overall Officials: David Delmonico, PhD, Study Director — Chair of the Duquesne University IRB
Locations (4):
- United States (4):
  - Pioneer Hospital, Brawley, California
  - El Centro Regional Medical Center, El Centro, California
  - University of California, San Diego, San Diego, California
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://drive.google.com/open?id=1vNjwT5j9Y32e7vdayZAMBp-3PvJWCiSK